CLINICAL TRIAL: NCT00002438
Title: Randomized Study Comparing Itraconazole to Placebo in the Prevention of Histoplasmosis in Patients With Human Immunodeficiency Virus Infection
Brief Title: A Study of Itraconazole in the Prevention of Histoplasmosis, a Fungal Infection, in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 235B; MSG 28; ITR-USA-73
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: HIV Infections; Histoplasmosis
Keywords: Itraconazole; Histoplasmosis; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Histoplasmosis; Acquired Immunodeficiency Syndrome | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
To assess the safety and efficacy of itraconazole versus placebo for prevention of histoplasmosis in HIV-infected patients with CD4 counts < 150 cells/mm3 who reside where histoplasmosis is endemic. To assess the safety and efficacy of itraconazole for preventing other debilitating fungal infections, such as cryptococcosis, aspergillosis, recalcitrant oropharyngeal or vaginal candidiasis, and recurrent esophageal candidiasis.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Residence in an area endemic for H. capsulatum.
* Absolute CD4 count < 150 cells/mm3.
* No current or past active histoplasmosis.
* No other active fungal infection.
* Life expectancy of at least 1 year.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Life-threatening infection or malignancy other than cutaneous Kaposi's sarcoma.
* Inability to take oral medication.

Concurrent Medication:

Excluded:

* Systemically-active antifungals.
* Investigational drugs (expanded access drugs are acceptable).
* Rifampin.
* Rifabutin.
* Terfenadine.
* Astemizole.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.
* H2 blockers.
* Omeprazole.
* Continual antacids.

Patients with the following prior conditions are excluded:

History of intolerance to imidazole or azole compounds.

Prior Medication:

Excluded within 1 month prior to study entry:

* Investigational drugs (expanded access drugs are acceptable).

Excluded within 15 days prior to study entry:

* Rifampin.
* Rifabutin.
* Terfenadine.
* Astemizole.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Infectious Diseases of Indianapolis, Indianapolis, Indiana
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Infectious Diseases Association / Research Med Ctr, Kansas City, Missouri
  - ASCC, Memphis, Tennessee
  - Dr Michael Threikeld, Memphis, Tennessee
  - Dr Mark A Pierce, Nashville, Tennessee